CLINICAL TRIAL: NCT04123483
Title: EnBrace HR for Premenstrual Syndrome (PMS) With Prominent Mood Symptoms (or Menstrual Related Mood Disorders, MRMD)
Brief Title: EnBrace HR for PMS With Prominent Mood Symptoms or Menstrual Related Mood Disorders
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Cancellation of funding contract
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Marlene P. Freeman, Associate Director, Center for Women's Mental Health, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2019P002454
Record Dates: First submitted 2019-10-09; First posted 2019-10-11 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Premenstrual Syndrome; Premenstrual Dysphoric Disorder; Premenstrual Tension; Menstrual Related Mood Disorder
Keywords: PMS; Folate; Omega-3 Fatty Acids; Vitamins; Women's Health; Dietary Supplements; PMDD; MRMD; Menstrual Related Mood Disorder; Premenstrual Tension
MeSH Terms: conditions — Premenstrual Syndrome; Premenstrual Dysphoric Disorder

STUDY DESIGN:
Intervention Model Description: A pilot study of EnBrace HR in a single group of women who experience PMS with prominent mood symptoms or a menstrual related mood disorder (MRMD). All women will be experiencing clinically significant menstrual related mood symptoms at the time of enrollment. In this study, EnBrace HR is studied for acute treatment PMS with prominent mood symptoms and MRMD.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- EnBrace HR for Acute Treatment of PMS and MRMD (Experimental): Prescription folate prenatal supplement with other dietary ingredients; one multiphasic soft gelatin capsule 1x/day for 8 weeks. Participants are currently experiencing clinically significant MRMD symptoms, defined as a ≥ 30% increase in the total Daily Record of Severity of Problems Scale (DRSP) score from the mid-follicular phase (average of DRSP scores for days 6-10) to the late-luteal phase (average of DRSP scores for last 5 days prior to menstrual bleeding).
  Interventions: Drug: EnBrace HR Softgel

INTERVENTIONS:
Drug: EnBrace HR Softgel — Prescription folate prenatal supplement with other dietary ingredients; one multiphasic soft gelatin capsule 1x/day for 8 week study
  Other Names: EnBrace HR

SUMMARY:
The purpose of this study is to assess a novel nutritional supplement developed for prenatal health and mood benefits, and to determine whether there is preliminary evidence for efficacy in Menstrual Related Mood Disorders (MRMD), including PMS with Prominent Mood Symptoms and PMDD.

DETAILED DESCRIPTION:
The luteal phase of the menstrual cycle, also referred to as the premenstrual phase, is a time of vulnerability for women, during which many suffer from a number of physical and psychiatric symptoms. Premenstrual mood symptoms affect a great proportion of women, and can affect general wellbeing, self-esteem, occupational and social functioning, and relationships. A spectrum of severity exists around the manifestation of these symptoms, and a range of terms can be used to refer to women with substantial psychiatric morbidity around the luteal phase of the menstrual cycle.

Premenstrual Dysphoric Disorder (PMDD) has been formalized as a psychiatric diagnosis and added to the DSM-5. For a diagnosis of PMDD, the diagnostic criteria include the following and must be met for most menstrual cycles in the preceding year: A) In the majority of cycles, at least five symptoms must be present in the final week before the onset of menses and start to improve within a few days of its onset, B) One or more of the following must be present: 1) affective lability, 2) irritability/anger or increased interpersonal conflicts, 3) depressed mood, hopelessness or self-deprecating thoughts, 4) anxiety or tension. Also, one or more of the following must be present: 1) decreased interest in usual activities, 2) difficulty concentrating, 3) low energy or fatigue, 4) change in appetite or cravings, 5) increased or decreased sleep, 6) feeling overwhelmed or out of control, 7) physical symptoms (i.e., breast tenderness, bloating, weight gain).

Several overlapping definitions and terms capture psychiatric distress related to the luteal phase of the menstrual cycle. Many women suffer substantially during the premenstrual phase but do not have symptoms that fully meet criteria for PMDD. The term menstrual related mood disorder (MRMD) has been used to describe conditions that include Premenstrual Dysphoric Disorder (PMDD) and also mood dysregulation related to the menstrual cycle that is clinically substantial but where the threshold for a PMDD formal diagnosis is not met. Premenstrual Syndrome (PMS) refers to recurrent premenstrual symptoms that may include mood symptoms, but mood symptoms may not be present in all women with PMS.Therefore, a subset of women with PMS with prominent (or marked) mood symptoms would be included under the category of MRMD. Therefore, in addition to those who meet full criteria for PMDD, many women suffer from premenstrual syndrome (PMS) with prominent mood symptoms. The term menstrual related mood disorder (MRMD), applies to women who may or may not meet the threshold for the formal PMDD diagnoses and represents a great number of women of reproductive age who suffer on a regular basis from luteal phase mood symptoms that compromise quality of life.

Previous pre-clinical or clinical studies leading up to and supporting the research The prevalence of PMDD is between 3-8% of menstruating women; in addition, another 10-11% experience PMS with Prominent Mood Symptoms.1 Based on these estimates, 13-19% of menstruating women experience MRMD, including those with both PMDD and PMS with prominent mood symptoms, on a consistent basis.

Menstrual related mood disorders (MRMDs) are characterized by prominent symptoms during the luteal phase of the cycle, with relief starting with the onset of menses or soon after menses start. The follicular phase is generally asymptomatic, and the difference in symptom expression between worsening during the luteal phase and improvement during the follicular phase is its hallmark. While many women recognize these patterns of cyclic mood worsening and the impact upon quality of life, many women do not seek treatment. For women who do seek treatment from health care providers, the first line pharmacologic treatments are serotonergic antidepressants and oral contraceptive pills. For women who prefer other options, such as complementary and alternative medicine treatments or nutritional approaches, few treatments have received rigorous study. There is some promising but limited research with integrative treatments, such as light therapy, supplements, and herbal treatments.

Objective: To evaluate the efficacy of EnBrace HR when used to treat premenstrual syndromes (PMS) with predominant mood symptoms, also referred to as MRMD.

Specific Aim 1: To evaluate the effect of treatment with EnBrace HR in women with prominent mood symptoms in the premenstrual phase of the menstrual cycle. EnBrace will be administered in a continuous daily regimen, and the outcome will be the effect on the mean DRSP during the luteal phase from baseline to the treatment cycle 1 and 2 assessments.

Exploratory Aims: To evaluate the effect of EnBrace HR with respect to:

1. Mean change from baseline to endpoint in CGI-S scores
2. Tolerability and safety
3. To assess whether biomarkers can be identified that appear to be associated with treatment response to EnBrace HR

The current study will provide evidence regarding the efficacy, tolerability, feasibility and acceptability of a selected non-psychotropic treatment alternative to serotonergic antidepressants and oral contraceptive pills. We hypothesize that the prevalence of PMDD, MRMD, and PMS in menstruating women may be attenuated if there are other effective treatments available to women.

ELIGIBILITY:
Inclusion Criteria:

1. Regular menstrual cycles, 23-35 days in length.
2. MRMD diagnosis based on the DRSP items, with: at least 1 or more core symptoms occurring during the luteal phase of the menstrual cycle for at least the past three months by patient history, including: 1) low mood, 2) hopelessness, 3) feeling worthless or guilty, 4) feeling anxious or "keyed up" or "on edge," 5) mood swings, 6) more sensitive to rejection or to hurt feelings, 7) feeling angry/irritable, or 8) having interpersonal conflicts.
3. Patients must also have at least 1 associated symptom on the DRSP that is not considered a core symptom that occurs during the luteal/premenstrual phase of the menstrual cycle.
4. Currently experiencing clinically significant MRMD symptoms, defined as ≥ 30% increase in the total Daily Record of Severity of Problems Scale (DRSP) score from the mid-follicular phase (average of DRSP scores for days 6-10) to the late-luteal phase (average of DRSP scores for last 5 days prior to menstrual bleeding).
5. Negative serum Human Chorionic Gonadotropin (HCG) at baseline, and negative urine HCG at visits 3 and 5.
6. Willingness to use adequate contraceptive methods during the study, if sexually active. Hormonal contraceptives are allowed if the premenstrual symptoms still meet study criteria despite use and patient has been on a stable regimen for >3 months.
7. Good general health.

Exclusion Criteria:

1. Amenorrhea or irregular menstrual periods (defined as unable to predict within 7 days) during past 2 months.
2. Pregnant and lactating women.
3. Women taking a prenatal vitamin, methotrexate, fluorouracil, colchicine, bromocriptine, Gonadotropin-Releasing Hormone (GnRH) agonists, vitamin B6 (>100 mg), calcium supplements (>1500 mg per day), or para-aminosalicylic acid.
4. Significant risk for self-harm or harm to others.
5. Meet criteria for a primary diagnosis of schizophrenia, bipolar disorder, an active eating disorder of anorexia or bulimia, dementia, delirium, or other cognitive disorder.
6. Current major depressive episode or anxiety disorder that is a primary focus of current treatment. Patients may be on an antidepressant used for maintenance treatment if the dose is not changed intermittently to address premenstrual symptoms; dose must be stable for at least 8 weeks prior to study entry.
7. Presence of an active substance and/or alcohol abuse disorder within six months prior to screening.
8. Known low B12 levels, pPernicious anemia or history of gastric bypass surgery or bariatric surgery.
9. Seizure disorder or current use of an anticonvulsant medication
10. Allergy to beeswax, soy, fish, nuts, peanuts, egg, wheat, milk, and/or shellfish.
11. Non-English speaking.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-11 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Rate of Treatment Response to EnBrace Therapy Measured Using The Daily Record of Severity of Problems (DRSP) | Assessed daily for 8 weeks of treatment
  Experience a response (50% improvement in MRMD symptoms) to EnBrace therapy, as assessed by the DRSP (≥ 50% decrease in DRSP score during the luteal phase). The DSRP involves daily rating of scale items and ranking based on severity for each day of the menstrual cycle. The DRSP includes 21 symptom items grouped within 11 domains. An individual records the score for each item on each day using the following scale of 1 to 6: 1=not at all, 2=minimal, 3=mild, 4=moderate, 5=severe, 6=extreme. Clinically significant MRMD symptoms are defined as a ≥ 30% increase in the total DRSP score from the mid-follicular phase (average of DRSP scores for days 6-10) to the late-luteal phase (average of DRSP scores for last 5 days prior to menstrual bleeding).

CONTACTS AND LOCATIONS:
Overall Officials: Marlene P Freeman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No